CLINICAL TRIAL: NCT04781361
Title: Comparison of the Effects of Isotonic and Hypotonic Intravenous Maintenance Fluids on Term Neonatal Babies Undergoing Intravenous Fluid Therapy: Multicenter Observational Neofluid Study
Brief Title: Comparison of the Isotonic and Hypotonic Intravenous Maintenance Fluids In Term Newborns: Neofluid Study
Acronym: NEOFLUID
Status: Completed | Type: Observational
Sponsor: Dokuz Eylul University (Other)
Collaborators: Izmir Katip Celebi University (Other); Dr. Behcet Uz Children's Hospital (Other); Eskisehir Osmangazi University (Other); Necmettin Erbakan University (Other); NCR International Hospital (Unknown); Uşak University (Other); Zekai Tahir Burak Women's Health Research and Education Hospital (Other); Aydin Adnan Menderes University (Other); Inonu University (Other); Baskent University (Other); Kecioren Education and Training Hospital (Other); Istanbul University (Other); Istanbul Medeniyet University (Other); Dr. Lutfi Kirdar Kartal Training and Research Hospital (Other Government); Kanuni Sultan Suleyman Training and Research Hospital (Other); Medipol University (Other); Cukurova University (Other); Mersin Training and Research Hospital (Other Government); Cigli Regional Training Hospital (Other); Gulhane School of Medicine (Other); Ministry of Health University, Bursa Yüksek İhtisas Training and Research Hospital (Unknown); Yuksek Ihtisas University (Other); Ministry of Health University, Kayseri Regional Hospital (Unknown); Suleyman Demirel University (Other); Konya Private Medova Hospital (Unknown); Ankara Yildirim Beyazıt University (Other); Cumhuriyet University (Other); Aydın Maternity and Children Hospital (Unknown); Umraniye Education and Research Hospital (Other Government); Selcuk University (Other); Mersin University (Other); Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Funda Tuzun, M.D., Associate Professor of Neonatology, Dokuz Eylul University
Other Study IDs: 363-SBKAEK
Record Dates: First submitted 2021-02-04; First posted 2021-03-04 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Newborn Complication; Hyponatremia of Newborn; Hypernatremia of Newborn; Fluid Therapy; Sodium Chloride; Isotonic Dehydration
Keywords: Newborn, fluid therapy, isotonic, hypotonic,NaCl
MeSH Terms: interventions — Glucose

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Isotonic fluid: Group, received isotonic maintenance fluid containing NaCl between 131 to 154 mmol/L such as:
  * Dextrose 5% in 0.9% NaCl,
  * Intravenous fluid containing NaCl between 131 to 154 mmol/L
  Interventions: Drug: Intravenous isotonic fluid - NaCl 131-154 mmol/L in 5% dextrose
- Hypotonic fluid: Group, received hypotonic maintenance fluid containing NaCl < 130 mmol/L such as:
  * Dextrose 5 % in 0.02 % NaCl,
  * Dextrose 5% in 0.033 % NaCl
  * Dextrose 5% in 0.045 % NaCl
  * Intravenous fluid containing NaCl < 130 mmol/L
  Interventions: Drug: Intravenous Hypotonic fluid- Sodium Chloride < 130 mmol/L

INTERVENTIONS:
Drug: Intravenous isotonic fluid - NaCl 131-154 mmol/L in 5% dextrose — Isotonic group will be given fluids containing 131-154 mmol/L Sodium Chloride
  Other Names: B05BB02, 0.9% NaCl/Dextrose 5%
  Groups: Isotonic fluid
Drug: Intravenous Hypotonic fluid- Sodium Chloride < 130 mmol/L — Hypotonic group will be given fluids containing lower than 130 mmol/L :
  Dextrose 5% in 0.2% Sodium Chloride, or Dextrose 5% in 0.33 % Sodium Chloride,or Dextrose 5% in %0.45 Sodium Chloride, or Intravenous fluid containing Sodium Chloride < 130 mmol/L
  Other Names: B05BB02, 0.45% NaCl/5% dextrose; B05BB02, 0.33 % NaCl/5% dextrose; B05BB02, 0.20 % NaCl/5% dextrose
  Groups: Hypotonic fluid

SUMMARY:
Considering the physiological changes in fluid and electrolyte balance and providing proper support are one of the important aspects of neonatal intensive care. Maintenance intravenous fluids are designed to maintain homeostasis when a patient is unable to uptake required water, electrolytes, and energy. Hypotonic fluids are still the most commonly prescribed IV fluids for pediatric hospitalized patients. However, previous studies, including children older than one month of age revealed that traditionally used hypotonic fluids may lead to hyponatremia.

Because of the absence of evidence-based data, there is currently no clear consensus on the optimal composition of maintenance intravenous fluid therapy in newborns, leading to wide practice variation.

The National Clinical Guideline Center (NICE) 2015 recommends the use of isotonic fluids in term newborn infants and some newborn centers has begun to use isotonic fluids since guidelines recommendations. Since the publication of the NICE guideline, no studies have addressed this topic.

In this prospective, observational , multicentric study, conventional hypotonic fluids containing sodium chloride (NaCl) < 130 mmol/L compared with isotonic fluids (containing NaCl between 131-154 mmol/L) in terms of the risk of hyponatremia, hypernatremia, plasma sodium (pNa) level change, treatment morbidities, hospitalization duration and mortality.

ELIGIBILITY:
Inclusion Criteria are:

* Term newborns (>37 + 0/7 weeks) aged 24 hours to 30 days with a normal baseline serum sodium level between 135-145 mmol/L,with a treatment plan to include IV fluids at > 50% of maintenance
* Infants not received parenteral fluids in the last 24 hours before participation
* Infants receiving IV fluid administration at 50% to 100% of maintenance

Exclusion Criteria:

* Newborns with diagnoses that required specific fluid tonicity and volumes such as:

  * Severe dehydration presenting with shock
  * Syndrome of inappropriate antidiuretic hormone secretion (SIADH)
  * Renal insufficiency
  * Adrenal insufficiency
  * Diabetes mellitus and diabetes insipidus
  * Hypoxic ischemic encephalopathy
  * Major congenital anomaly
  * Patients receiving diuretic therapy
  * Patients with obvious edema
  * Heart or liver failure, portal hypertension with acid
  * Pre-post operative patients
  * Infants receiving total parenteral nutritional therapy
  * Other: all conditions that require non-standard liquid content and quantities

Ages: 1 Day to 30 Days | Sex: All
Age Groups: Child
Study Population: Hospitalized term newborns (>37 weeks) , requiring iv fluid treatment after 24 hour postnatal age
Sampling Method: Probability Sample
Enrollment: 420 (Actual)
Dates: Start 2020-12-30 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Change in mean plasma Na | 24 hours after the intervention
  Change in mean plasma sodium levels per hour (∆pNa mmol/L/hour)
Rate of development of hyponatremia | during the intervention
  Plasma sodium (pNa) level <135 mmol/L
Rate of development of hypernatremia | during the intervention
  Plasma sodium (pNa) level >145 mmol/L

SECONDARY OUTCOMES:
Weight in kilograms | during the intervention
  weight gain
length of stay | during the intervention
  hospitalisation day
mortality | during the intervention
  mortality due to complications of administered fluid

CONTACTS AND LOCATIONS:
Overall Officials: Hasan Ozkan, Prof., Principal Investigator — Dokuz Eylül University- Faculty of Medicine
Locations (1):
- Dokuz Eylul University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] National Clinical Guideline Centre. IV Fluids in Children: Intravenous Fluid Therapy in Children and Young People in Hospital. London: National Institute for Health and Care Excellence (UK); 2015 Dec. Available from http://www.ncbi.nlm.nih.gov/books/NBK338141/ PMID 26741016
- [Background] Balasubramanian K, Kumar P, Saini SS, Attri SV, Dutta S. Isotonic versus hypotonic fluid supplementation in term neonates with severe hyperbilirubinemia - a double-blind, randomized, controlled trial. Acta Paediatr. 2012 Mar;101(3):236-41. doi: 10.1111/j.1651-2227.2011.02508.x. Epub 2011 Nov 19. PMID 22040311
- [Background] McNab S, Ware RS, Neville KA, Choong K, Coulthard MG, Duke T, Davidson A, Dorofaeff T. Isotonic versus hypotonic solutions for maintenance intravenous fluid administration in children. Cochrane Database Syst Rev. 2014 Dec 18;2014(12):CD009457. doi: 10.1002/14651858.CD009457.pub2. PMID 25519949
- [Background] Tuzun F, Akcura Y, Duman N, Ozkan H. Comparison of isotonic and hypotonic intravenous fluids in term newborns: is it time to quit hypotonic fluids. J Matern Fetal Neonatal Med. 2022 Jan;35(2):356-361. doi: 10.1080/14767058.2020.1718094. Epub 2020 Mar 29. PMID 32223482